CLINICAL TRIAL: NCT03228225
Title: Tele - Cardiac Rehabilitation - Providing Secondary Prevention and Supervised Exercise Without Boundaries of Time and Space - PILOT 1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Robert Klempfner Heart Rehabilitation Institute, Director of Cardiac rehabilitation institute, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMC-17-4154
Record Dates: First submitted 2017-07-17; First posted 2017-07-24 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: single arm non-blinded remote monitored multidisciplinary secondary prevention intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tele cardiac rehabilitation (Experimental): Following a standard intake process, patients will begin exercise in the institute and will gradually over a period of 6 months reduce the number of institution visits and will concomitantly increase the number of home \ community exercise sessions. During the entire period we will monitor program, coach and fine-tune the exercise program. Weekly exercise data will be securely transmitted to the rehabilitation team (heart rate zones, duration of exercise and type, step count, caloric expenditure, blood pressure and patients reported impressions)
  Interventions: Behavioral: Tele Cardiac Rehabilitation

INTERVENTIONS:
Behavioral: Tele Cardiac Rehabilitation — Comprehensive intervention according to the secondary prevention goals

SUMMARY:
We aim to enroll subjects eligible to cardiac rehabilitation that are defined as low-risk according to national guidelines. We plan to gradually reduce the number of institution based CR and increase the tele monitored exercise sessions performed in the community. Stress test will be preformed before the intervention and after completing 6 month.

DETAILED DESCRIPTION:
Following the standard rehabilitation intake process (physician visit, nurse intake, exercise physiologist consultation based on stress test and clinical data passed from the physician) all subjects will begin their secondary prevention program including on-site supervised training, nurse case management, plus dietitian and psychological consultation as necessary. During the study weeks subjects will wear the smartwatch (Polar Inc.) in order to collect de-identified data (heart rate, step count, walk speed etc.) and will upload data to the Polar cloud. No medical data will be uploaded and subjects will only have a coded ID randomly generated. During the exercise periods (both on-site in the cardiac rehabilitation institute, and also during the recommended community exercise performed on their own).

Gradually, the number of on-site sessions will decrease from the standard of 8 sessions per month to zero (each month after the first a reduction of 2 sessions). We plan to reduce the on-site sessions while increasing the number of home-based session in order to evaluate the ability to monitor, coach and dynamically adjust the exercise program by combined use of smartwatch data and telephone contact. Polar exercise watch will be provided and appropriate operation instructions and education will be given after informed consent.

During the 6 month study period we will contact subjects once or twice weekly in order to encourage participation, fine-tune the exercise program and to assess secondary prevention goals.

All subjects will undergo a stress test before and after 6 months of training part of the standard of care management, as well as dietitian, physician and psychologist consultations will be offered following the regular schedule of the standard rehabilitation program (at baseline, 3 months and 6 months).

ELIGIBILITY:
Inclusion Criteria:

* Coronary disease (S/p ACS, PCI, CABG or stable angina with documented coronary disease)
* Age ≥ 21
* Smartphone with internet connection
* Willing and able to comply with study protocol and
* LVEF > 40% and Baseline METS ≥ 5
* Able to follow the personalized exercise prescription, utilize smartwatch and upload exercise data per protocol

Exclusion Criteria:

* Heart failure (clinical) or unresolved significant arrhythmia (i.e. symptomatic atrial fibrillation)
* Significant neurological or cognitive impairment
* Women of child-bearing potential
* Symptomatic hypotension, orthostatic hypotension or repeated blood pressure systolic value <100 mmHg without symptoms
* ACS or percutaneous coronary intervention (PCI) within 30 days prior to screening, or having undergone CABG surgery within 30 days prior to screening
* Inability to perform a CPET test due to physical limitations
* Ischemia per stress test \ nuclear scan or stress echocardiography
* Severe angina pectoris as defined by CCS >2
* Pulmonary disease of severity greater than mild (COPD, Asthma, ILD, CTD with lung involvement) or chronic pulmonary thromboembolic disease (CTED)
* Severe orthopedic limitations
* Active myocarditis, constrictive pericarditis, restrictive or hypertrophic cardiomyopathy
* Moderate or severe Aortic or Mitral stenosis, moderate or severe mitral regurgitation due to primary valvular disease
* Significant anemia (Hb <10 mg/dl)
* Known drug or alcohol dependence or any other factors which will interfere with the study conduct or interpretation of the results or in the opinion of the investigator are not suitable to participate;

Any illness which reduces life expectancy to less than 1 year from screening

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-07-20 (Estimated); Study Completion 2018-08-01 (Estimated)

PRIMARY OUTCOMES:
Exercise capacity | 6 months
  Stress bases METS assessment

SECONDARY OUTCOMES:
Subject satisfaction | 3 and 6 months
  Questioner based assessment of program
Adherence to exercise program | 3 and 6 months
  Amount of time exercising at the specified target heart rate zone per week
Quality of life | 3 and 6 months
  QOL questioners
Device ease of use and technical difficulties | 1, 3 and 6 months
  Questioners and transmission failures or usability issues

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Undecided